CLINICAL TRIAL: NCT03598023
Title: A Randomized Clinical Investigation to Evaluate the Efficacy of Cytal® Burn Matrix in the Management of Partial-Thickness Burns to the Hand
Brief Title: A Study to Evaluate the Efficacy of Cytal® Burn Matrix in the Management of Partial-Thickness Burns to the Hand
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor discretion
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR2017-001
Record Dates: First submitted 2018-05-21; First posted 2018-07-26 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Partial Thickness Burn of Hand
Keywords: ACell; Hand; Burn; ACell Cytal Burn Matrix®; Extracellular Matrix; Urinary Bladder Matrix; Wound; Partial-Thickness; Burn Management
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Single-site, randomized, prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Active Comparator): Cytal® Burn Matrix
  Interventions: Device: Cytal® Burn Matrix
- Group 2 (Active Comparator): EZ-Derm® Porcine Xenograft
  Interventions: Device: EZ-Derm® Porcine Xenograft

INTERVENTIONS:
Device: Cytal® Burn Matrix — Cytal® Burn Matrix
  Arms: Group 1
Device: EZ-Derm® Porcine Xenograft — EZ-Derm® Porcine Xenograft
  Arms: Group 2

SUMMARY:
This is a randomized controlled trial (RCT) aimed at determining if use of Cytal® Burn Matrix in the management of partial-thickness burns to the hand shows improved wound healing times when compared to EZ-Derm Porcine Xenograft.

DETAILED DESCRIPTION:
A single site, two arm, parallel-design randomized trial comparing Cytal® Burn Matrix to EZ-Derm® Porcine Xenograft, for patients with partial-thickness burns to the hand. Up to 60 patients from a single center will be recruited and randomized (using a 1:1 randomization scheme) to receive either Cytal® Burn Matrix or EZ-Derm®. Scar formation, number of wounds requiring autografting, wound infections, rate of healing, hand function and impact of treatment will be compared between study arms. Additionally, a cost analysis and review of individual and group changes in narcotic prescription patterns and employment status will be evaluated. The protocol defined patient follow-up is 6 months.

An independent biostatistician will review all participant data for power and futility analysis. In addition, a clinical events committee will adjudicate adverse events (AEs) and serious adverse events (SAEs)

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female, 18 to 75 years of age.
2. Negative pregnancy test required.
3. Presence of partial thickness burns to one or both hands.
4. Thermal burn etiology.

Exclusion Criteria:

1. Allergy or hypersensitivity to materials in porcine-based study products or personal preference.
2. Friction, chemical, or electric burn etiology.
3. Immunosuppression.
4. Presence of a local and/or systemic infection.
5. Received prior treatment to the study site within 60 days of Screening.
6. Concurrent participation in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Complete Wound Healing | 6 months
  To Compare the time to complete wound healing between Groups 1 and 2

SECONDARY OUTCOMES:
Evaluation of Scar Formation | 6 months
  To assess, measure, and evaluate scar formation between Groups 1 and Group 2 using Vancouver Scar Scale (VSS). VSS is a scale from 0 (normal) to 13 on an index scale measuring pigmentation, pliability, height, vascularity, pain and pruritus.
Wounds Requiring Autografting | 6 months
  The total number of wounds that required the use of autografting by 6 months will be compared between Groups 1 and 2.
Wound Infections | 21 days
  The total number of burn wound infections between Group 1 and 2
Rate of Healing | 6 months
  Measured by change in wound surface area over time, in cm2/week between Groups 1 and 2.
Hand Function | 6 months
  Hand function measured by Michigan Hand Scale, Quick DASH and occupational therapy evaluation
  MHQ measures overall hand function, activities of daily living, pain, work performance, aesthetics, and satisfaction. The score ranges from 0 (worst) to 100 (best) performances and satisfaction. Pain ranges from 0(no pain) to 100 (worst pain).
  Quick DASH uses a 5 point Likert scale with 0(no disability) to 5(most severe disability) to measure disability/symptom and sport/music performance or work modules.
Impact of Treatment | 6 months
  Pain assessment using Visual Analog Pain Scale (VAS) and inpatient length of stay. VAS measures subjective characteristics or attitudes regarding perceived pain levels from participants. Participants are asked to draw a vertical line on a 10 cm horizontal line indicating what their current pain level would be with 0 being no pain and 10 being the worst pain imaginable. The distance between the start of the horizontal line to the vertical line is calculated in cm.
Compare treatment-emergent adverse event safety profile between Group 1 and Group 2 | 6 months
  Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Device Effects (UADEs) between Group 1 and 2. AEs being any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related. SAEs being any suspected adverse reaction considered "serious" by the Investigator or Sponsor. UADEs being any serious adverse effect associated with the device that affects the rights, safety, or welfare of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Blair Summitt, MD, Principal Investigator — Vanderbilt University Medical Center, Regional Burn Center; Wesley Thayer, MD, Principal Investigator — Vanderbilt University Medical Center, Regional Burn Center